CLINICAL TRIAL: NCT05733741
Title: Preservative-free Topical Anesthetics for the Management of Postoperative Pain Following Photorefractive Keratectomy
Brief Title: Preservative-free Topical Anesthetics for Post-PRK Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Abdel-Radi, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PFTAPRK
Record Dates: First submitted 2023-01-30; First posted 2023-02-17 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Myopia
Keywords: Post-PRK pain; Preservative-free topical anesthetics; Single-step PRK
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preservative-free topical anesthetics group (Experimental): Patients in this group had the standard post-PRK treatment regimen in addition to the prescription of preservative-free topical anesthetics for pain control following single-step transepithelial PRK surgery in one eye.
  Interventions: Drug: Preservative-free Benoxinate hydrochloride 0.4% (Benoxidia unit-dose vials [UD], Orchidia pharmaceutical Ind., Egypt)
- Preservative-free artificial tears group (Placebo Comparator): Patients in this group had the standard post-PRK treatment regimen in addition to the prescription of preservative-free artificial tears as a placebo following single-step transepithelial PRK surgery in the other eye.
  Interventions: Drug: Preservative-free Sodium hyaluronate 0.2% (Polyfresh unit-dose vials [UD], Orchidia pharmaceutical Ind., Egypt).

INTERVENTIONS:
Drug: Preservative-free Benoxinate hydrochloride 0.4% (Benoxidia unit-dose vials [UD], Orchidia pharmaceutical Ind., Egypt) — For each patient, one eye was treated with preservative-free Benoxinate hydrochloride 0.4%.
  The prescribed regimen comprises of the instillation of one drop immediately, 2, 4, 6 and 8 hours after the end of surgery.
  Every patient was given 5 UD vials only of preservative-free Benoxinate hydrochloride 0.4% at each follow up visit for the next postoperative day usage administered 5 times daily (every 3 hours while awake) for the first 3 postoperative days giving clear instructions to immediately discard the vial after single use.
  Arms: Preservative-free topical anesthetics group
Drug: Preservative-free Sodium hyaluronate 0.2% (Polyfresh unit-dose vials [UD], Orchidia pharmaceutical Ind., Egypt). — The other eye was treated with preservative-free Sodium hyaluronate 0.2%. The prescribed regimen comprises of the instillation of one drop immediately, 2, 4, 6 and 8 hours after the end of surgery.
  Every patient was given 5 UD vials only of preservative-free Sodium hyaluronate 0.2% at each follow up visit for the next postoperative day usage administered 5 times daily (every 3 hours while awake) for the first 3 postoperative days giving clear instructions to immediately discard the vial after single use.
  Arms: Preservative-free artificial tears group

SUMMARY:
The goal of this interventional comparative study is to assess the efficacy and safety of a novel regimen of preservative-free unit-dose topical anesthetics for controlling early postoperative pain following single-step transepithelial PRK surgery.

The main research questions to answer are:

* Question 1: Are topical anesthetics effective in reducing post-PRK pain?
* Question 2: Are short-term topical anesthetics toxic to the cornea?
* Question 3: How to prevent abuse of topical anesthetics by patients at home?

Participants were planned to undergo a bilateral single-step transepithelial PRK surgery to correct their refractive errors and received a standard post-PRK treatment regimen for both eyes. Additionally, one eye was offered a preservative-free topical anesthetic as an experimental group and the other eye was offered a preservative-free artificial tear as a control group.

DETAILED DESCRIPTION:
Photorefractive keratectomy (PRK) is a well-established surface ablation procedure for correction of refractive errors which involves the removal of corneal epithelium in a large diameter usually more than 6 mm followed by stromal ablation.

Early postoperative pain within the first few days after surgery is one of the commonest complications reported after PRK. The classic postoperative treatment includes the prescription of topical antibiotics and frequent preservative-free lubricants to accelerate epithelial healing.

The current treatment regimens also includes topical steroids, topical non-steroidal anti-inflammatory drugs (NSAID) and oral NSAID to reduce inflammation and post-PRK pain.

Earlier studies suggested that topical anesthetics in diluted concentrations and fractional doses didn't delay corneal epithelial regeneration after PRK but their use didn't gain popularity because of problems with topical formulation, stability and preservation.

ELIGIBILITY:
Inclusion Criteria:

Patients who are candidate for PRK surgery with

1. Myopia up to - 6 diopters or myopic astigmatism up to - 4 diopters.
2. Corneal thinnest pachymetry of 500 µm
3. Residual stromal bed more than 350 µm after epithelial ablation.

Exclusion Criteria:

Patients with

1. Corneal scars or dry eye disease,
2. Past ocular surgery,
3. History of contact lens wear,
4. Systemic diseases such as diabetes mellitus and autoimmune diseases,
5. History of oral analgesics abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Postoperative pain score on the verbal rating scale (VRS) | 1 week
  The doctor asks the patient to choose the word that best describes his/her pain and then gives it a score from zero to 4 (Zero for no pain, 1 for mild pain, 2 for moderate pain, 3 for severe pain and 4 for unbearable pain).
Postoperative pain score on the visual analogue scale (VAS) | 1 week
  The patient is asked to rate his/her pain by choosing a number on a scale from zero to 10 considering zero as no pain and 10 as worst possible pain.

SECONDARY OUTCOMES:
Corneal epithelial healing duration | 1 week
  Time for the corneal epithelium to heal reported in days after PRK surgery
Endothelial cell density (ECD) | from preoperative to 1 month postoperative.
  Specular microscopy was used to assess endothelial cell count before and after PRK surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Abdel-Radi, MD, Principal Investigator — Assiut University
Locations (1):
- Tiba Eye Center, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Steigleman WA, Rose-Nussbaumer J, Al-Mohtaseb Z, Santhiago MR, Lin CC, Pantanelli SM, Kim SJ, Schallhorn JM. Management of Pain after Photorefractive Keratectomy: A Report by the American Academy of Ophthalmology. Ophthalmology. 2023 Jan;130(1):87-98. doi: 10.1016/j.ophtha.2022.07.028. Epub 2022 Oct 4. PMID 36207168
- [Derived] Abdel-Radi M, Eldaly Z, Alattar S, Goda I. Preservative-Free Topical Anesthetic Unit-Dose Eye Drops for the Management of Postoperative Pain Following Photorefractive Keratectomy. Ophthalmol Ther. 2023 Dec;12(6):3025-3038. doi: 10.1007/s40123-023-00791-0. Epub 2023 Sep 4. PMID 37665497